CLINICAL TRIAL: NCT02785627
Title: Assessment of Bone Loss in Men Receiving Treatment for Prostate Cancer
Acronym: ANTELOPE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Prof Janet Brown (Other)
Collaborators: Sheffield Teaching Hospitals NHS Foundation Trust (Other); Weston Park Hospital Cancer Charity (Other)
Responsible Party: Sponsor-Investigator, Prof Janet Brown, Professor of Translational Medical Oncology, University of Sheffield
Organization: University of Sheffield (Other)
Other Study IDs: STH18645
Record Dates: First submitted 2016-05-19; First posted 2016-05-30 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Prostate Cancer
Keywords: Bone health; Bone microarchitecture; Androgen deprivation therapy (ADT)
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group A: ADT: Men with non-metastatic prostate cancer, about to start or within 2 weeks of starting ADT
  Interventions: Other: Comprehensive bone health assessment
- Group B: ADT + chemotherapy: Men with newly diagnosed hormone sensitive metastatic prostate cancer, starting ADT and who will have chemotherapy
  Interventions: Other: Comprehensive bone health assessment
- Group C: Controls: Healthy age matched men
  Interventions: Other: Comprehensive bone health assessment

INTERVENTIONS:
Other: Comprehensive bone health assessment — Blood sample taken for biomarkers of bone turnover, anthropometric measurements, assessments of physical function, DXA scan, HR CT T12 vertebra, Xtreme pQCT radius

SUMMARY:
The ANTELOPE trial is a longitudinal observational clinical study of changes in bone density, structure and strength over 12 months in men receiving treatment for prostate cancer. Three groups (n = 30 per group) will be compared, with bone assessments at baseline and 12 months. Allowing for a 18 month recruitment period, 12 months follow-up and data analysis, the total study length will be 3 years. The groups comprise:

Group A - Men with prostate cancer starting ADT

Group B - Men with newly diagnosed hormone sensitive metastatic prostate cancer, about to start (or have started within the past 3 months) ADT and who will undergo chemotherapy with docetaxel and prednisolone

Group C - Age-matched men without prostate cancer

DETAILED DESCRIPTION:
Prostate cancer is the commonest non-skin cancer in men, with more than 40,000 new cases diagnosed in the UK each year. Development of prostate cancer depends upon testosterone (the male hormone), and medications that block testosterone (eg Androgen Deprivation Therapy, ADT) can help men to survive for many years. Men with metastatic prostate cancer are also treated with ADT, but recent evidence has demonstrated that there are survival benefits when chemotherapy given as well as ADT. Many patients now receive chemotherapy as first line treatment along with ADT in the context of newly diagnosed metastatic disease.

However, blocking testosterone causes bone loss which may lead to osteoporosis and increases the risk of osteoporotic fracture. Such fractures cause pain, loss of mobility and independence, and one in three men who have a hip fracture will die within one year. The osteoporosis caused by prostate cancer treatments may differ from other forms; the limited available data suggest that it may affect the wrist more than other bones (most other forms affect the spine and hip the most). We need to better understand the pattern of osteoporosis in these men, so that we can offer the most effective treatment to protect their bones and ensure that they stay as well as possible as they live with their cancer treatment

The aim of this study is to determine the effect of prostate cancer treatment on bone health. Comprehensive bone assessment at baseline and 12 months will include different bone scans (DXA whole body, Xtreme CT of radius and HR CT T12 vertebra), biochemical markers of bone turnover, anthropometric measurements, and assessment of grip strength and muscle strength and function.

ELIGIBILITY:
Inclusion Criteria:

All participants

* Men aged 50-80 years old, WHO performance status ≤2.
* Have provided written informed consent prior to any trial-specific procedures
* Able and willing to comply with the terms of the protocol and to undertake the trial assessments
* Body Mass Index (kg/m2) >18.5 and <35.0
* No evidence of significantly abnormal organ function on standard laboratory testing

Group A

* Histological confirmation of prostate cancer
* No indication of metastatic disease
* Scheduled to commence ADT (but must have baseline assessments carried out within 4 weeks of commencement of ADT). Those starting ADT are expecting to have a duration of treatment of 12 months or more.
* No prior systemic therapy for advanced prostate cancer (not receiving concurrent anti-neoplastic therapy, besides ADT or an anti-androgens), participants may have received radiotherapy or may receive this during the study period

Group B

* Men with newly diagnosed hormone sensitive metastatic prostate cancer who have commenced ADT and who have been referred for chemotherapy
* Bone metastases will be allowed provided not in the radius (DXA measurement will attempt to image sites with no/minimal bone metastases)
* Men who have received palliative radiotherapy for known bone metastases prior to or during the study may be included, but the site of radiotherapy must be accurately recorded and attempts will be made to avoid such sites in subsequent DXA measurement.
* Men with bone pain due to known bone metastases may receive necessary analgaesia, including opiates, as needed on study
* Participants in group B will be allowed to continue oral corticosteroids, provided that the dose does not exceed 2mg dexamethasone or 10 mg prednisolone daily. Men in this group may also receive additional steroids as prophylaxis during chemotherapy.

Group C

• Men that do not have a diagnosis of prostate cancer

Exclusion Criteria:

* Known metabolic bone disease or other diseases (other than prostate cancer) known to affect bone metabolism including: hyperthyroidism, primary hyperparathyroidism, chronic liver disease, rheumatoid arthritis, inflammatory bowel disease or malabsorption

  * Medications (in addition to ADT) known to affect bone metabolism including osteoporosis treatments and anti-epileptics
  * Previous hormone treatments within 1 month (other than ADT in Groups A and B)
  * Any concurrent or recent other invasive cancer that could confuse diagnosis or endpoints. Allowed situations include, but are not limited to, non-melanoma skin cancer, superficial bladder cancer (if in doubt please discuss with trial team).
  * Fracture or orthopaedic surgery within the last 12 months
  * Arthritis, orthopaedic surgery or other abnormality of the radius, spine or hip which would prevent accurate acquisition of study measurements.
  * Current or prior (within one month) participation in any other clinical trial involving a medicinal product, except STAMPEDE for men in group B. For other trial, please consult trial team.
  * For Group B, those on bisphosphonates or alpha-radon on study entry are excluded (but please see separate advice on Pg 19 for men who need to go on bisphosphonates or alpha-radon whilst on study).
  * Groups A and C: Men taking oral systemic corticosteroids (inhaled steroids will be permitted). In Group B oral corticosteroids are permitted, provided that the dose does not exceed 2mg dexamethasone or 10mg prednisolone daily. Those in group B may also receive additional steroids given as prophylaxis alongside chemotherapy

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men aged 50-80 years
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-03 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Change in volumetric bone mineral density at the distal radius | 12 months
  Assessed by HR-pQCT in the ADT group (Group A)and compared to the control group (Group C)

SECONDARY OUTCOMES:
Characterisation of the microstructural pattern of bone loss in men receiving treatments for prostate cancer. | 12 months
  This will be assessed by HR-pQCT of the distal radius, which gives detailed information regarding the bone volume ratio, trabecular number, derived trabecular thickness, derived trabecular separation, and volumetric bone mineral density. These will be compared in men receiving ADT/chemotherapy and compared with age-matched healthy controls and cortical thickness
Correlation of bone loss and microstructural change with biochemical markers of bone turnover, serum testosterone levels and changes in muscle strength and body composition. | 12 months
  Determining whether bone loss and changes in bone microarchitecture are associated with changes in biomarkers of bone turnover measured in the serum, and changes in strength and body composition
Characterisation of the microstructural pattern of bone loss at the spine (T12) | 12 months
  A comparison of bone loss and changes in bone microarchitecture at the T12 vertebra using HRCT in men receiving treatments for prostate cancer compared with age-matched, healthy controls

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Clinical Trials Centre, Sheffield, South Yorkshire, United Kingdom